CLINICAL TRIAL: NCT03411746
Title: Evaluation of New Neuroinflammation Markers in Subarachnoid Haemorrhage Patients: a Pilot Study
Brief Title: Evaluation of the Level and Prognostic Relevance of New Neuroinflammation Markers in Subarachnoid Haemorrhage
Acronym: ESA-MICROPN
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Rosanna Vaschetto, MD, PhD, Prof., Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE 115/17
Record Dates: First submitted 2018-01-04; First posted 2018-01-26 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum, urine, liquor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Subarachnoid haemorrhage — Data on the type of patients enrolled have been described already in other sections.

SUMMARY:
Subarachnoid hemorrhage (SAH) consists of blood extravasation into the space between arachnoid and pia mater. Bleeding is a consequence of cerebral aneurysm rupture in most cases. Despite incidence being only 9 cases out of 1000 people per year, young age and high mortality and morbidity lead to loosing several years of healthy life. Therapy priorities are: preventing rebleeding, with endovascular treatment (when possible) or neurosurgical aneurism clipping; preventing complications associated with blood extravasation into subarachnoid pace, such as acute hydrocephalus treatment (that occurs in 20% of patients), by ventricular external drainage positioning, and delayed cerebral ischemia, mainly due to vasospasm, by endovenous administration of nimodipine; optimal perfusion pressure maintenance.

Endogenous osteopontin (OPN) is thought to fulfill a protective activity over ischemic damage both in brain and other organs, including kidney. Besides, recombinant OPN administration markedly decreases ischemic area in a focal cerebral ischemia model, by an antiapoptotic action. Recent in vivo studies on animal models of SAH demonstrated that OPN plays a major role: treatment with OPN seems to prevent vasospasm reducing smooth muscle cells and endothelial cells apoptosis.

Microparticles are mediators released by platelets, leucocytes, erythrocyte and endothelial cells. In ischemic stroke endothelial microparticles levels directly relate to clinical severity and ischemic area extension. In typical parenchymal haemorrhage microparticles levels are higher both in blood and in liquor and associated with worse clinical outcome. In SAH increased microparticle levels have been demonstrated, especially in the days of the bleeding, and microparticle levels change based on subtypes. Data disagree about the subtypes involved and their time course. This study aims to evaluate the correlation between OPN and microparticles levels and vasospasm development/ischemic lesion at the CT-scan, and subsequently with medium and long-term patients outcome.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) consists of blood extravasation into the space between arachnoid and pia mater. Bleeding is a consequence of cerebral aneurysm rupture in most cases. It particularly affects females with an average age of 55 years. Despite incidence being only 9 cases out of 1000 people per year, young age and high mortality and morbidity lead to loosing several years of healthy life. As a matter of fact, patients that survived cerebral aneurysm rupture suffer from cognitive deficits, behavior disorders and are unable to come back to their former productivity level and jobs. Therapy priorities are: preventing rebleeding, with endovascular treatment (when possible) or neurosurgical aneurism clipping; preventing complications associated with blood extravasation into subarachnoid pace, such as acute hydrocephalus treatment (that occurs in 20% of patients), by ventricular external drainage positioning, and delayed cerebral ischemia, mainly due to vasospasm, by endovenous administration of nimodipine; optimal perfusion pressure maintenance. Under a pathophysiological point of view, after early mechanical damage, caused by aneurysm rupture (due to tissue destruction consequent to hemorrhage mass effect, acute hydrocephalus, herniation or a possible intraparenchymal hematoma) a subacute damage could be developed from three to fourteen days post haemorrhage, because of delayed cerebral ischemia. Mainly responsible for this event are vasospasm, that complicates 20-30% of SAH, microcirculation dysfunction and microthromboembolism. Secondary damage pathogenesis is not clear, but inflammation and endothelial apoptosis are shown to be involved in vasospasm development. Moreover, some studies demonstrate that patients with acute neurological dysfunction have a grater risk of organ failure, especially for lungs and kidneys.

Osteopontin (OPN) is a secreted extracellular matrix glycoprotein that plays several roles in physiological and pathological processes, such as tissue remodelling, fibrosis, cellular migration, apoptosis inhibition and inflammation. Endogenous OPN is thought to fulfil a protective activity over ischemic damage both in brain and other organs, including kidney. Besides, recombinant OPN administration markedly decreases ischemic area in a focal cerebral ischemia model, by an antiapoptotic action. Recent in vivo studies on animal models of SAH demonstrated that OPN plays a major role; its administration attenuates cerebral damage decreasing metalloproteinase 9 and inhibiting inducible nitric oxide synthase. Treatment with OPN seems to prevent vasospasm as well, inducing an endogenous mitogen-activated protein (MAP) inhibitor, i.e. MAP kinase phosphatase 1, and reducing smooth muscle cells and endothelial cells apoptosis. A further research field in this area concerns microparticles, that is mediators released by platelets, leucocytes, erythrocyte and endothelial cells. Contrary to what it used to be thought, they do not represent a form of waste material from apoptotic coagulation cells and recent studies show their paracrine ad regulatory activity. In ischemic stroke endothelial microparticles levels directly relate to clinical severity and ischemic area extension. In typical parenchymal haemorrhage microparticles levels are higher both in blood and in liquor and associated with worse clinical outcome. In SAH increased microparticles levels has been demonstrated, especially in the day of the bleeding, and microparticles levels change based on type. On the other hand, data disagree among papers about types involved in fluctuations and their time course: Lackner et al. evaluated 20 SAH patients (Fisher II, III and IV) in their first fifteen days from bleeding and found higher blood levels of platelet, endothelial, erythrocyte and leukocyte microparticles in comparison to healthy controls [28]. Moreover, endothelial type positive for cluster of differentiation (CD) 105 and CD 62 markers were particularly increased in patient affected by vasospasm, documented with doppler. Vasospasm associated ischemia, also present especially high levels of platelet CD 41 positive microparticles. Notwithstanding disability grade at the time of discharge, microparticles levels are higher in comparison to full recovered patients (n=11). More recently, Sanborn et al. study on 22 SAH patients with massive blood spreading (Fisher III and IV) confirms microparticles elevation levels in these patients. Elevation of endothelial and platelet microparticles levels is verified as well, while no correlation is found with evidence of vasospasm, in both ultrasound (mean velocity higher than 125 cm/s in anterior circulation or higher than100 cm/s in posterior circulation, in addition to a Lindegaard ratio higher than 3) and angiography.

Published data are not unanimous on neither the correlation between vasospasm and CT scan evidence of ischemia nor with disability.

The primary endpoint of the study is to evaluate:

1) the correlation between OPN and microparticles levels and vasospasm development/ischemic lesion at the CT-scan, and subsequently with medium and long-term patients outcome.

Secondary endpoints were:

1. Changings of OPN amount in liquor and blood of patients with SAH on the day of bleeding and post-hemorrhage i.e., days 1, 2, 3, 5, 7, 9, 11.
2. Microparticles levels in liquor and blood patients with SAH on the day of bleeding and post hemorrhage i.e., days 1, 2, 3, 5, 7, 9, 11, in order to evaluate both their predictive value for vasospasm and the correlation with renal or pulmonary function worsening and 3-6 months outcome.
3. Isolated microparticles will be used to activate in vitro renal and pulmonary endothelial cells for the purpose of highlighting a possible cross talk, analyzing endothelial damage markers.

Recruitment duration will be one year. At hospital entry, a CT scan will be performed as well as Fischer score, Hunt and Hess score and World Federation of Neurological Surgeons (WFNS) score. We will register demographic variables i.e., age, sex, symptoms at onset and co-morbidity.

Angiography or angio-CT scan will be performed according to the best clinical practice to document presence, dimension and characteristics of patent aneurysm. SAH patients' treatment will be carried out as routine clinical best practice. Patients will be monitored with transcranial doppler beginning from day I and clinically every day. If no clinical changing will occur, patients will be submitted to a CT perfusion angiography or angiography on day 7 (+/- 1 day). If clinical condition worsen or doppler velocity increase (considering vasospasm as mild when mean velocity inside cerebral artery 120-150 cm/s, moderate 150-200 cm/s and severe >200 cm/s) angiography and endovascular nimodipine will be considered, according to the standard protocol therapy. Angiographic vasospasm consists in cerebral arteries narrowing confirmed by neuroradiologist. Clinical vasospasm is defined as consciousness deterioration (Glasgow coma scale (GCS) 2 points reduction) and/or a new focal deficit emergence, after other causes has been excluded, such as seizure, rebleeding, fever. Every new CT evidence of ischemia will be registered from day 3.

At 3-6 months outcome will be evaluated by GOS-E (Extended Glasgow Coma Scale; 8 points scale, from death to upper good recovery, without any disability left related to SAH). To obtain this information, trained staff will interview either patients himself or a close relative.

Biological samples will be taken at admission, i.e., within 24 hours from the bleeding, and in days 1, 2, 3, 5, 7, 9, 11. Sterile liquor will be sampled from the bag distal to collection chamber, in an amount of 10 ml/die, at the same time frame each day. Blood in amount of 3 ml/die and urine will be collected at the same time (about 7:00 am). Liquor, plasma and urine will be centrifuge (2500 rpm for 30 minutes) and supernatants will be aliquoted and frozen at the temperature of -80°C until analysis. OPN analysis will be performed with commercial enzyme-linked immunosorbent assay (ELISA) kit, following manufacturer suggestion (AssayDesigns Inc., Michigan; Pierce Biotechnology Inc., Rockford, IL). In order to better describe inflammatory response, main T helper 1 (Th)1 and Th2 cytokines will be measured as well as cerebral damage markers (enolase neuron specific (NSE), asymmetric dimethylarginine (ADMA) etc.). On urine, markers of early preclinical impairment will be quantified. Isolation and characterization of microparticles will be performed with Nanosight based on dimension and concentration, while major surface antigens will be identified in cytofluorimetry, specifying provenience: leukocyte, erythrocyte, platelet, endothelial cells. In vitro analysis will be carried out on renal and pulmonary endothelial cells monolayer. Water balance, creatinine, leukocytes number, infection/colonization, nephrotoxic drugs will be monitored daily.

Microparticles effect will be evaluated in vitro on umbilical cord endothelial cells (HUVEC), on smooth muscle cells (SMC), on pulmonary and renal endothelial cells, incubated with and without patients' plasma derived purified microparticles. In addition, analysis will be performed to evaluate: apoptosis (Tunel staining), angiogenesis (evidence of capillary-like structures on Matrigen plate), leukocyte adhesion and adhesion molecule expression.

As no data are present in literature on OPN levels during SAH and data on microparticles are not unanimous, a real sample size was not calculated. Considering that 20%-30% of the patients were expected to be complicated with vasospasm, the enrollment was planned with 60 patients in one year to get 12-18 patients with vasospasm. Participants matching inclusion and exclusion criteria will be enrolled both in ICU and Neurosurgery Ward of Novara Ospedale Maggiore della Carità in one year period (i.e. January 31 st 2018, January 30 th 2019). Based on last year admissions, 20 patients in ICU and 40 patients in Neurosurgery ward are expected. At T0, microparticles levels will be analyzed in patients with and without vasospasm with Wilcoxon rank test. With generalized steam equations microparticles levels will be compared between patients with and without vasospasm or new ischemic events. 3 and 6 months GOS-E will be compared using Kruskal-Wallis test. The relation between microparticles number and vasospasm and ischemia incidence will be defined with Spearman correlation. A value of p less than 0.05 will be the threshold for statistical significance. Analysis will be carried out with STATA. As far as concerns in vitro experiments, non-parametric tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Subarachnoid haemorrhage from cerebral aneurysm rupture
* Indication to external liquor drainage

Exclusion Criteria:

* Age less than 18 or more than 80 years
* Bleeding occurred more than 24 hours before admission
* Known coagulopathies or antiplatelet or vitamin K antagonist treatment

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid haemorrhage admitted to Neurosurgery or ICU of Ospedale Maggiore della Carita will be considered eligible, when meeting including criteria, within 24h from bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation between OPN and microparticle levels and vasospasm development/ischemic lesion at the CT-scan, and subsequently with medium and long-term patients outcome. | Day 7 is the day expected for cerebral vasospasm. Therefore for the correlation between OPN/microparticles and vasospasm/ischemic lesion at CT scan will be evaluated on day 7.
  The levels of OPN and microparticles will be related to:
  1. the presence or absence of vasospasm development
  2. the presence or absence of ischemic lesion at the CT-scan
  3. 3-6 months outcome evaluated with the GOS-E

SECONDARY OUTCOMES:
In vitro stimulation of renal and pulmonary endothelial cells with microparticles | Microparticles isolated from patient blood on the day of the expected maximum release, i.e., day 7 will be incubated in vitro with renal and pulmonary endothelial cells.
  Isolated microparticles will be used to activate in vitro renal and pulmonary endothelial cells for the purpose of highlighting a possible cross talk, analyzing endothelial damage markers.

OTHER OUTCOMES:
Levels of OPN in liquor and blood of patients with SAH | Time course of OPN levels measured the day of bleeding and on days 1, 2, 3, 5, 7, 9, 11.
  Increase compared to the baseline i.e., day of the bleeding, of OPN level in liquor and blood of patients with SAH measured on days 1, 2, 3, 5, 7, 9, 11.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Vaschetto, Professor, Principal Investigator — Università degli Studi del Piemonte Orientale Amedeo Avogadro
Locations (1):
- Rosanna Vaschetto, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou C, Yamaguchi M, Colohan AR, Zhang JH. Role of p53 and apoptosis in cerebral vasospasm after experimental subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2005 May;25(5):572-82. doi: 10.1038/sj.jcbfm.9600069. PMID 15729295
- [Background] Schroeter M, Zickler P, Denhardt DT, Hartung HP, Jander S. Increased thalamic neurodegeneration following ischaemic cortical stroke in osteopontin-deficient mice. Brain. 2006 Jun;129(Pt 6):1426-37. doi: 10.1093/brain/awl094. Epub 2006 Apr 24. PMID 16636021
- [Background] Huang M, Hu YY, Dong XQ. High concentrations of procoagulant microparticles in the cerebrospinal fluid and peripheral blood of patients with acute basal ganglia hemorrhage are associated with poor outcome. Surg Neurol. 2009 Nov;72(5):481-9; discussion 489. doi: 10.1016/j.surneu.2008.12.016. Epub 2009 Mar 27. PMID 19328537
- [Background] Sanborn MR, Thom SR, Bohman LE, Stein SC, Levine JM, Milovanova T, Maloney-Wilensky E, Frangos S, Kumar MA. Temporal dynamics of microparticle elevation following subarachnoid hemorrhage. J Neurosurg. 2012 Sep;117(3):579-86. doi: 10.3171/2012.6.JNS111163. Epub 2012 Jul 13. PMID 22794324